CLINICAL TRIAL: NCT05356260
Title: URincontrol4men: Self-management Through an App, Compared to the Consultation of a General Practitioner for Men With Lower Urinary Tract Symptoms
Brief Title: Self-management Compared to Care-as-usual for Men With Lower Urinary Tract Symptoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Bekkenbodem4All (Unknown); Leiden University Medical Center (Other); University of Twente (Other); Isala (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZonMW 852002125
Record Dates: First submitted 2022-04-01; First posted 2022-05-02 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower urinary tract symptoms; eHealth; Self-management; Primary care
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Pragmatic non-inferiority randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (Active Comparator): CAU will be that typically provided by GPs. Also patients will be informed about a page on thuisarts.nl regarding male LUTS. The pragmatic trial design means that care can vary depending on the preferences of patients and GPs in this group.
  Interventions: Other: Care as usual
- Online self-management intervention (Experimental): Participants in the intervention group will be given access to an online self-management program that will be personalized. This program was developed based on the results of a literature search, the opinions of expert Dutch GPs and urologists, and a pilot study in secondary care, with further preliminary testing in primary care. The program consists of nine components: information, pelvic floor exercises, bladder training, sitting voiding position, urethral milking, fluid management, caffeine avoidance, alcohol avoidance, and physical activity increase. Information is presented as text with supportive figures, plus audio (a "read aloud function" for all text) and video fragments to facilitate engagement by men with low literacy levels.
  Interventions: Device: URincontrol4men

INTERVENTIONS:
Device: URincontrol4men — The intervention is built as an app
  Arms: Online self-management intervention
Other: Care as usual — CAU will be that typically provided by GPs. Also patients will be informed about a page on thuisarts.nl regarding male LUTS. The pragmatic trial design means that care can vary depending on the preferences of patients and GPs in this group.
  Arms: Care as usual

SUMMARY:
Research question: Does offering an online self-management program lead to more efficient use of care by men with urinary complaints? Hypothesis: Many men with urinary symptoms receive medication from their GP. Advice on how to self-manage complaints is often skipped. This while self-management is effective. By offering self-management instead of visiting a GP the use of care by men with urinary complaints may decrease and treatment may become more efficient.

Study design: Men are randomized to receive either care-as-usual by their GP or the online self-management program. Men will be followed for six months and the cost-effectiveness of the online self-management intervention will be compared to the care-as-usual

DETAILED DESCRIPTION:
Rationale: Although self-management can be difficult to implement because it is time consuming to explain, it has proven effective for LUTS. For this reason, we developed an online intervention that can be used at home by men with LUTS, giving tailored advice to each case. Objective: To assess the effectiveness and cost-effectiveness of providing an online personalized self-management program as a first-line intervention to men with lower urinary tract symptoms (LUTS) compared to care as usual (CAU).

Study design: A pragmatic non-inferiority randomized controlled trial in the general population. Study population: Men with LUTS (>18 years of age) who are considering visiting a general practitioner for their complaints.

Intervention: Access to an online program offering personalized selfmanagement advice compared to care as usual Main endpoints: Outcomes will be assessed at 6 weeks, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Men with lower urinary tract symptoms who are thinking about visiting a GP for their complaints

Exclusion Criteria:

* Men with complicated LUTS who should seek urgent care, including those with nocturnal incontinence (e.g., chronic urinary retention), the inability to void despite urgency (e.g., acute urinary retention), and with sudden onset or worsening LUTS (e.g., urinary tract infections).
* Men receiving treatment from a pelvic physiotherapist, GP, or urologist (including at any point in the previous year).
* Men with a history of prostate cancer, bladder cancer, or urinary tract surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
The Patient Global Impression of Improvement (PGI-I) | 6 months
  The PGII is a single-question global index for change of incontinence symptoms that is rated with a 7-point Likert scale ranging from "very much worse" to "very much better." This variable will be dichotomized into "improved" (scores ≥ "better") and "not improved."

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire Male Lower Urinary Tract Symptoms Module (ICIQ-MLUTS) | 6 weeks and 6 months
  The ICIQ-MLUTS is a questionnaire for evaluating male lower urinary tract symptoms and impact on quality of life. Its has two subscales; voiding symptoms (range 0 -20) and incontinence symptoms (range 0-24) with higher scores indicating more symptoms.
International Prostate Symptom Score Quality of Life (IPSS QoL) | 6 weeks and 6 months
  International Prostate Symptom Score (single item) quality of life. The score ranges from 0 - 6 with a higher score indicating a lower quality of life.
the EuroQol instrument (EQ-5D-5L) | 6 weeks and 6 months
  The EQ-5D-5L is s generic quality of life questionnaire. Utilities can be calculated from this questionnaire with a maximum score of 1 indicating a perfect health state.
iMTA Medical Consumption Questionnaire (iMCQ) | 6 months
  Costs of medical consumption
iMTA Productivity Cost Questionnaire (iPCQ) | 6 months
  Costs of productivity losses

CONTACTS AND LOCATIONS:
Overall Officials: Marco Blanker, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The processed, anonymised data will be made available in DataverseNL and a persistent identifier to a minimal dataset(s) will be given in the publication(s).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publishing of the manuscripts related to this study
Access Criteria: Requests for re-use of data will be evaluated by the Principal Investigator who will check whether the research question falls within the scope of the informed consent. There will be terms and conditions drawn up in a contract for re-using data by third parties.